CLINICAL TRIAL: NCT03937869
Title: A Multi-Center, Open-Label Study to Evaluate the Safety of a Single Oral Dose of Solosec™ (Secnidazole) 2g Oral Granules for the Treatment of Adolescent Girls With Bacterial Vaginosis
Brief Title: Evaluate the Safety of a Single Oral Dose of Solosec™ (Secnidazole) 2g for the Treatment of Adolescent Girls With BV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lupin Research Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYM-1219-401
Record Dates: First submitted 2019-04-22; First posted 2019-05-06 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Bacterial Vaginoses
Keywords: Adolescents; Vaginal fishy smell; Vaginal itching; off-white milky vaginal discharge
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — secnidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose Solosec (secnidazole) 2g oral (Other): Solosec 2 grams, oral
  Interventions: Drug: Secnidazole

INTERVENTIONS:
Drug: Secnidazole — One dose
  Other Names: Solosec™

SUMMARY:
A multi-center, open-label study to evaluate the treatment of one oral dose of 2g Solosec™ (Secnidazole) in adolescent girls with BV

DETAILED DESCRIPTION:
This is a multi-center, open-label study to evaluate the safety of Solosec in adolescent girls with bacterial vaginosis. Approximately 40 patients will be enrolled. Patients determined to be eligible at the Baseline Visit (Day 1) will receive a single oral dose of Solosec™ granules (containing 2 grams of secnidazole) on Day 1. Patients will return to the site once between Days 7-14 for a "test of cure" (TOC) Visit. A follow-up telephone call will be performed at Days 21-30 to assess the continued clinical response to treatment and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Are adolescent girls 12-17 years of age.
2. Are willing and able to give written informed assent with a written informed consent from a parent or legal guardian. (Amendment 01- Assent only if State allowed)
3. Are in good general health including as confirmed by a medical history and physical examination, with no known medical or mental health conditions that, in the Investigator's opinion, may interfere with study participation.
4. Willing and able to participate in the study as an outpatient, make required visits to the study center, and comply with all study requirements.
5. Have a negative urine pregnancy test result prior to study treatment initiation. In addition, female patients of childbearing potential must be using an acceptable form of birth control as determined by the Investigator (e.g., oral contraception, implantable, injectable or transdermal hormonal contraception, intrauterine device [IUD], double-barrier methods, have a vasectomized partner or abstinence [if the patient becomes sexually active they must use one of the acceptable methods of birth control]). Note: NuvaRing® or any other vaginal ring products are not permitted.
6. Have a clinical diagnosis of bacterial vaginosis, defined as having all of the following criteria:

   1. Off-white (milky or gray), thin, homogeneous vaginal discharge AND
   2. Vaginal pH > 4.5 AND
   3. Presence of Clue cells of ≥ 20% of the total epithelial cells on microscopic examination of the vaginal saline wet mount AND
   4. A positive 10% KOH Whiff test.
7. Agree to abstain from vaginal intercourse until after the TOC visit.
8. Agree not to have any vaginal penetration or use of any vaginal products until after the TOC visit (e.g., spermicides, condoms, diaphragms, vibrators, tampons, etc.).
9. Agree not to use vaginal douches or similar products for the duration of the study.

Exclusion Criteria:

1. Are pregnant, lactating, or planning to become pregnant during the study.
2. Are menstruating or have vaginal bleeding at the Baseline Visit (Day 1).
3. Are menopausal as determined by the Investigator.
4. Are suspected clinically (or confirmed diagnostically) of having alternative causes of vaginal symptoms including candidiasis, Chlamydia trachomatis, Trichomonas vaginalis, Neisseria gonorrhoeae or Herpes simplex or human papilloma virus.
5. Have active genital lesions, including active Herpes simplex lesions, or other vaginal or vulvar conditions which could confound the interpretation of the clinical response, as determined by the Investigator (patients with genital warts that are not being treated may be enrolled).
6. Have received antifungal or antimicrobial therapy (systemic or intravaginal) within 14 days prior to the Baseline Visit (Day 1).
7. Are using NuvaRing® or any other vaginal ring products.
8. Have consumed any alcohol within 12 hours prior to treatment with study medication.
9. Have a history of drug or alcohol abuse within the past 6 months, as determined by the Investigator.
10. Have participated in any investigational trial within 30 days or six half-lives of the test drug's biologic activity, whichever is longer, before the Baseline Visit (Day 1).
11. Are participating in any investigational, observational or non-interventional study (either currently or during the study).
12. Have had previous exposure to SYM-1219 or participation in other clinical trials of SYM-1219.
13. Have a known allergy to nitroimidazoles (e.g., metronidazole, tinidazole, nimorazole, etc.).
14. Have a history of an abnormal Pap smear which required cervical biopsy or cervical cauterization within 3 months of the Baseline Visit (Day 1).
15. Have any history of cervical carcinoma or other carcinomas of the vagina or vulva.
16. Have any condition that interferes with their ability to understand or comply with the requirements of the study.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — must be adolescent females ages 12-17 years of age
Enrollment: 40 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome Responder | At TOC visit study day 7-14
  Defined as patients with resolution of abnormal vaginal , negative 10% KOF WHIFF test, and Clue cells less than 20% of the total epithelial cells
Nugent Score | At TOC visit study day 7-14
  All patients with a score of 0-3 will be considered normal; scores of 4 and above will considered abnormal.
Investigator Clinical Assessment | At TOC visit study day 7-14
  Investigator's opinion of the need for additional BV treatment. (Yes/No)
Patient's Continued Clinical Response | At TOC visit study day 7-14
  Investigator's opinion of the continued clinical response to treatment (Yes/No)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Site 1004 - Investigational Research Center, Long Beach, California
  - Site 1005 - Investigational Research Center, Hialeah, Florida
  - Site 1001 - Investigational Research Center, Miami Lakes, Florida
  - Site 1010 - Investigational Research Center, Sarasota, Florida
  - Site 1013, Tampa, Florida
  - Site 1011 - Investigational Research Center, Bardstown, Kentucky
  - Site 1008 - Investigational Research Center, Saginaw, Michigan
  - Site 1007 - Investigational Research Center, Memphis, Tennessee
  - Site 1006 - Investigational Research Center, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03937869/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03937869/SAP_001.pdf
  • Informed Consent Form (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03937869/ICF_002.pdf